CLINICAL TRIAL: NCT00128375
Title: Financial Incentives for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 802295; 1R01DP000100-03 (NIH)
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation; Work-site; Incentives; Cost Effectiveness; Health Behavior; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Health Behavior; Smoking

INTERVENTIONS:
Behavioral: Financial incentives

SUMMARY:
The purpose of this study is to test the effectiveness of financial incentives for increasing long-term smoking cessation rates among employees at General Electric worksites throughout the United States.

DETAILED DESCRIPTION:
Smoking is the leading cause of preventable mortality in United States, accounting for approximately 435,000 of the 2.4 million deaths each year in the United States. Most smokers make multiple attempts to quit smoking, but only 2-3% succeed each year. Smoking cessation programs have proven effective in helping smokers quit, but only about 5% of smokers enroll in smoking cessation programs each year.

Financial incentives have been shown to increase enrollment in smoking cessation programs and short-term quit rates, but have not been well tested as a mechanism for increasing long-term quit rates. The existing evidence suggests that they could be highly effective, particularly among heavy smokers and low income smokers. In addition, financial incentives for smoking cessation will likely be more cost effective than most covered health services and at least as cost effective as other recommended smoking cessation treatments.

This study is a two-arm randomized clinical trial of financial incentives for smoking cessation among a sample of 850 male and female smokers from GE Energy worksites throughout the U.S. Smokers will be randomized to receive either usual care (information about local community-based smoking cessation resources, coverage of prescription drugs and physician visits) or usual care plus a package of financial incentives that includes $100 for completion of a community-based tobacco cessation program, $250 for short-term smoking cessation at either 3 months or 6 months after randomization, and $400 for smoking cessation 6 months post-quit date (biochemically confirmed).

ELIGIBILITY:
Inclusion Criteria:

* Employees of General Electric at work sites in the United States
* Current smokers who report having smoked at least 5 cigarettes per day for the prior 12 months
* Age 18 or older

Exclusion Criteria:

* Current use of other tobacco products, such as chewing tobacco, pipes, or cigars
* Planning to leave General Electric within the next 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878
Dates: Start 2005-03; Study Completion 2008-04

PRIMARY OUTCOMES:
Biochemically verified smoking cessation rates at 6 months post-quit date

SECONDARY OUTCOMES:
Enrollment in and completion of community-based smoking cessation programs within the first 6 months after randomization
Short-term quit rates at 3 months or 6 months post-quit date
Quit rates at 12 months post-quit date

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Volpp, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683